CLINICAL TRIAL: NCT06053827
Title: Embryo Transfer in Natural vs Substituted Cycle and the Scheduling Pattern of IVF
Brief Title: Natural Frozen Embryo Transfer (FET) vs Substituted Frozen Embryo Transfer (FET)
Status: Completed | Type: Observational
Sponsor: Clinique Ovo (Industry)
Responsible Party: Sponsor
Other Study IDs: 3356
Record Dates: First submitted 2023-09-19; First posted 2023-09-26 (Actual); Last update posted 2025-12-09 (Actual); Status verified 2025-12

CONDITIONS: Fertility Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Frozen embryo transfer substituted cycle: In a substituted cycle, estrogen and progesterone are given and a transfer is planned when the endometrium is ready
  Interventions: Other: Frozen embryo transfer
- Frozen embryo transfer natural cycle: In a natural cycle no hormones are given and a transfer is planned when there is a dominant follicle apparent at the ultrasound
  Interventions: Other: Frozen embryo transfer

INTERVENTIONS:
Other: Frozen embryo transfer — A frozen embryo transfer involves thawing a fertilized embryo and transferring it in the uterus in order to obtain a pregnancy

SUMMARY:
In frozen embryo transfer substituted cycles, patients are treated with progesterone and estrogen in an attempt to mimic the natural cycle and a transfer is planned whenever the endometrium is ready. In contrast, in frozen embryo transfer natural cycle patients are not taking any hormones, only triggered with hCG (human chorionic gonadotropin) when a dominant follicle is ready or they wait for the disappearance of the dominant follicle to plan the transfer date. Some doctors and centres shift towards using the substituted protocol in an attempt to make scheduling easier with less frequent ultrasounds.

This study will aim to compare clinical and biochemical pregnancy rates in patients who underwent frozen embryo transfers in natural cycles vs substituted cycles at the centre.

ELIGIBILITY:
Inclusion Criteria:

* Age < 40 years old
* Women having undergone either a frozen embryo transfer in natural cycle or substituted cycle
* IVF and FET cycles done at Clinique OVO

Exclusion Criteria:

* egg or embryo recipient
* History of recurrent miscarriages, defined as ≥ 3 consecutive losses
* Patients that needed Viagra, Plasma-Rich Platelet (PRP) or other modalities to improve their endometrial thickness
* Uterine abnormalities
* Abnormal hormonal profiles
* FET Stimulated cycles
* History of recurrent implantation failure defined as failed ≥ 2 euploid embryos transfer or ≥ 3 blastocysts

Max Age: 40 Years | Sex: Female
Age Groups: Child, Adult
Gender Based: Yes — Women able to have an embryo transfered in their uterus
Study Population: Data spreadsheet from Jan 2022 to March 2023 of patients undergoing natural or substituted frozen embryo transfer
Sampling Method: Probability Sample
Enrollment: 1207 (Actual)
Dates: Start 2023-09-19 (Actual); Primary Completion 2023-11-30 (Actual); Study Completion 2024-07-18 (Actual)

PRIMARY OUTCOMES:
Evaluate the clinical pregnancy rate of embryo transfer in natural vs substituted cycles | 6 to 8 weeks after Frozen Embryo Transfer
  clinical pregnancy is the presence of fetal heartbeat at the viability ultrasound

CONTACTS AND LOCATIONS:
Overall Officials: Camille Sylvestre, MD, Principal Investigator — clinique ovo R&D department
Locations (1):
- Clinique Ovo, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No